CLINICAL TRIAL: NCT04127669
Title: Double-blind, Randomised, Placebo-controlled Study to Evaluate the Efficacy and Safety of OSU6162 in the Treatment of Residual Symptoms After Stroke
Brief Title: Study Evaluating Efficacy and Safety of OSU6162 in the Treatment of Residual Symptoms After Stroke
Acronym: OSU6162DB003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arvid Carlsson Research AB (Industry)
Collaborators: Gottfries Clinic AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSU6162DB003; 2016-003888-19 (EudraCT Number)
Record Dates: First submitted 2019-10-09; First posted 2019-10-15 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Stroke Sequelae
Keywords: residual symptoms; mental fatigue; dopamine stabilizer
MeSH Terms: conditions — Mental Fatigue | interventions — OSU 6162

STUDY DESIGN:
Intervention Model Description: This study is a randomised, placebo-controlled, parallel-group (two-armed) study of 16 weeks' treatment duration, comparing OSU6162 with placebo treatment in patients with residual symptoms after stroke.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization done externally. IMP codes are contained in sealed envelopes (one envelope for each randomized patient) locked in a drawer at the Gottfries Clinic AB. No envelope is opened prior to the end of the study unless it is critical for the treatment/outcome of an adverse event. In the event of a medical emergency, essential for the clinical management or welfare of the patient, the Investigator may decide to break a patient's treatment code. If the blind is broken, the Investigator must notify the monitor as soon as possible without revealing the patient's study treatment assignment, unless the information is important for the safety of the patients remaining in the study. The Investigator will record the date and reason for breaking the blind for that patient in the hospital records. The coded medicine packages are distributed to the site where the study nurse/investigator are responsible for dispensing the packages to the patients according to the randomization list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Active substance treatment with OSU6162. Starting dose for all patients in the OSU6162 treatment group is 15 mg BID. The dose is taken orally as one circular coated tablet of 15 mg together with a light meal in the morning and one tablet around lunch unless otherwise agreed upon. In order to aim at optimal dosing of OSU6162, some flexibility is allowed. The investigators are able to modify the dose for individual patients based on how well the treatment is tolerated and how well the patients respond to it. In the case where there is no clear response, the dose can be increased to maximally 30 mg BID (intermediate dosage is allowed) after 4 weeks of treatment; it is also possible to decrease the dose to a lower level (even below 15 mg BID) if a higher dose is not tolerated and/or there is a perceived weakened therapeutic effect with the higher dose. All dose changes will be performed while retaining the blind.
  Interventions: Drug: OSU 6162
- Arm B (Placebo Comparator): Placebo treatment. Starting dose for all patients in the placebo group is one circular coated tablet (with identical appearance to active treatment tablets 15 mg) taken BID, according to the same schedule as active treatment. The dose may be increased or decreased in the same manner as for active treatment.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: OSU 6162 — The active ingredient of OSU6162 is the S-enantiomer with the chemical name (S)-3-[3-(methylsulfonyl)phenyl]-1-propylpiperidine hydrochloride. The substance is a white powder with a melting point of 177-182°C. Solubility in water is > 2000 mg/ml. Current laboratory code used is OSU6162-HCl. In trial protocol, OSU6162-HCl is shortened to OSU6162.
  Other Names: OSU6162-HCl; PNU-9639 1A
  Arms: Arm A
Drug: Placebo oral tablet — Circular coated tablet (with identical appearance to active treatment tablets 15 mg).
  Arms: Arm B

SUMMARY:
Following stroke, a recovery process is promptly initiated, which leads to a partial rehabilitation. However, a number of disabling residual symptoms may persist for years and include mental fatigue, depression, cognitive deficits, neurological problems and more. In the lack of an effective treatment these symptoms will lead to major consequences for the individual and the surrounding society. OSU6162 has in earlier clinical studies of stroke patients shown evidence of a favorable effect on residual symptoms, especially mental fatigue, together with a mild side effect profile.

In this phase II, randomized, placebo-controlled, two-armed study, a 16 week OSU6162 treatment will be compared to an equally long placebo treatment in patients with residual symptoms following stroke.

DETAILED DESCRIPTION:
Main objectives of this study are to evaluate the efficacy and safety of OSU6162 compared to placebo with respect to treatment response in post stroke patients.

Endpoints:

Primary endpoint is Clinical Global Impression of Change (CGI-C) after 16 weeks of treatment.

Secondary endpoints are:

CGI-C score after 4, 8 and 12 weeks of treatment. FAI; MFS; FSS; BDI; SF-36 scores after 4, 8, 12 and 16 weeks of treatment. Correlation between plasma concentration of OSU6162 and therapeutic response after 4 and 16 weeks of treatment.

Safety variables: AE/SAE, physical and neurological examinations, vital signs (blood pressure and puls) and laboratory test.

Study Design:

The treatment period is 16 weeks, during which all patients will make 7 study visits and have 4 telephone interviews.

Study visits include:

Visit 1: screening at week -2, Days -14 to -5 Visit 2: baseline at week 0 Visit 4: week 4 ± 3 days Visit 6: week 8 ± 3 days Visit 8: week 12 ± 3 days Visit 10: week 16 ± 3 days Visit 11: follow up at week 20 ± 7 days

Randomization and start of treatment with OSU6162 or placebo at baseline, visit 2, week 0. Study medication administered during all study visits from baseline at visit 2 to visit 8 at week 12.

Physical and neurological examinations, vital signs and weight recording during all study visits.

ECG recorded during visits 1 (week -2) and 10 (week 16). Blood (and urine) sampling for safety labs during visits 1 (week -2), visit 4 (week 4), visit 10 (week 16). Pregnancy test at visit 1 and 10.

Blood sampling for analysis of plasma OSU6162 concentration at visit 4 and 10.

Primary outcome measures and secondary outcome self-assessment tests performed during all study visits.

Telephone interviews at visit: 3 (week 2 ± 3 days), 5 (week 6 ± 3 days), 7 (week 10 ± 3 days) and 9 (week 14 ± 3 days.

Concomitant medication, adverse events and drug compliance are recorded during all visits and telephone interviews.

Dosing:

All patients in the OSU6162 group start with a dose of 15 mg BID. The dose is increased to a maximum of 30 mg BID after 4 weeks of treatment. Intermediate doses are allowed and the final dose is individually flexible, depending on the therapeutic response and presence of AE. In the placebo group patients receive tablets with identical appearance to active treatment tablets (OSU6162 15 mg), administered according to the same dosing regime as active treatment.

Data analysis and statistics:

Efficacy analyses will be based on Mixed Models for Repeated Measures (MMRM) analyses. The MMRM analyses use all the longitudinal observations at each post-baseline visit for the study period of interest. Significance tests will be based on estimated population marginal means and Type III test of fixed effects, using a two-sided test with the significance level of 0.05. Differences in distributions of categorical variables will be tested using the Chi-square test or Fisher's exact test.

Due to the large number of variables engendered, multivariate statistical evaluations will be performed as a complement to the above-mentioned statistical methods.

Before unblinding of the study data, a separate Statistical Analysis Plan (SAP) will be prepared.

Patient and data safety:

This study is conducted in accordance with the study protocol, the Declaration of Helsinki, ICH E6 GCP, the European Clinical Trials Directive 2001/20/EC and applicable local laws and regulations.

The Investigator is responsible for ensuring the accuracy, completeness, legibility and timeliness of the data recorded in the CRFs. Data recorded in the CRF that are derived from source documents should be consistent with the source documents or the discrepancies should be explained. Signed sections of CRFs are monitored and collected on a regular basis.

An individual secrecy agreement is established for all Sponsor, site personnel, independent auditors, and representatives from Competent Authorities that will have access to the information in the medical records for the participating patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Between 18-80 years
3. Stroke >12 months prior to the start of the study. Patients must have had the location of their stroke evaluated through a CT scan, noted in their hospital notes
4. Anamnestic evidence of post stroke residual symptoms at least 3 months prior to the start of the study
5. At least 10.5 points on Mental Fatigue scale at the screening visit 1 (week -2)

Exclusion Criteria:

1. Residual symptoms following other pathologies than stroke
2. Active substance abuse (drug screen taken at visit1)
3. Other serious somatic or psychiatric disease
4. Beck Depression Inventory >30 at visit1 and 2
5. Current pregnancy or breast-feeding, or intention to become pregnant within 3 months after the last dose
6. Female patients of childbearing potential not using adequate contraceptives. Female patients of childbearing potential must, for inclusion, use a highly efficient method of contraception, i.e. a method with a failure rate of less than 1% (e.g. sterilisation, hormone implants, hormone injections, some intrauterine devices, or vasectomy in partner). Male patients must agree to use condoms during the study and for 2 weeks after the end of the study/last dose of IMP, unless their partner is using a highly efficient method of contraception, as described above.
7. Pathologic ECG, as assessed by the investigator. Max QTc time on ECG: 450 ms in men and 460 ms in women
8. Abnormal laboratory values of such severity that participation in the study, in the opinion of the investigator, is questionable
9. Patients who are so debilitated by their disease that they are not assumed to be able to perform the assessments or handle the instruments used for evaluation of effect
10. Current participation in other Clinical trials
11. Previous treatment with OSU6162
12. Clinically significant liver disease which may prevent the patient from completing the study and/or an elevation in either total bilirubin, alkaline phosphatase, AST, ALT of >2 times the laboratory reference
13. Clinically significant renal disease which may prevent the patient from completing the study and/or an elevation in serum creatinine of >1.5 times the laboratory reference.
14. Any surgical or medical condition which, in the opinion of the investigator, might interfere with the absorption, distribution, metabolism or excretion of OSU6162
15. Patients treated with Modiodal, Xyrem, Mirtazapine, Mianserin or metabolic enzyme inhibitors (with the exception of antidepressants other than Mirtazapine and Mianserin) or inducers, or drugs with a narrow treatment window (e.g. warfarin, antiepileptics, cyclosporine) and individually modelled drugs such as lithium.
16. Use of drugs capable of inducing hepatic enzyme metabolism (e.g., barbiturates, rifampicin, carbamazepine, phenytoin, primidone) within 30 days prior to the start of the study (or 5 half-lives of the inducing agent, whichever is longer)
17. Antipsychotic treatment
18. Patients treated with "unstable therapies", i.e., treatments that have not been at the same dose for at least 6 weeks prior to inclusion in this study. The treatment must also remain unchanged during the study period. Insomnia medication and other PRN medications are allowed
19. Use of acute or chronic medications for other medical conditions are allowed based on the investigator's judgement. Occasional use of over-the-counter (OTC) medication is allowed at the investigator's discretion
20. Supplements from health food stores and naturopathic preparations (dietary supplements, natural remedies) are not allowed during the course of the study or 4 weeks before study start.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression of Change (CGI-C) | Assessment at week 16
  The CGI-C is a 7-point scale that requires the clinician to assess how much the patient´s illness has improved or worsened relative to a baseline state at the beginning of the study. CGI-C is rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Rating is performed by interviewing the patient to assess function and mental status.

SECONDARY OUTCOMES:
Clinical Global Impression of Change (CGI-C) | Assessment at week 4, 8, and 12.
Change in Frenchay Activity Index (FAI) | Assessment at baseline and at week 4, 8, 12, and 16.
  Change in FAI score is studied by comparing baseline value with values at several assessment points throughout the study.
  FAI is a measure of instrumental activities of daily living for use with patients recovering from stroke. The FAI assesses a broad range of activities associated with everyday life. The index consists of 15 questions.
Change in Mental Fatigue Scale (MFS) | Assessment at baseline and at week 4, 8, 12, and 16.
  Change in MFS score is studied by comparing baseline value with values at several assessment points throughout the study.
  The MFS is a self-assessment questionnaire to investigate the therapeutic effects of OSU6162 with focus on the mental fatigue and concentration capacity.
  The scale consists of 15 items of which 13 measure mental symptoms. Either reduced or increased sleep is measured. Variations around the clock are also rated.
Change in Fatigue Severity Scale (FSS) | Assessment at baseline and at week 4, 8, 12, and 16.
  Change in FSS score is studied by comparing baseline value with values at several assessment points throughout the study.
  The FSS is a 9-item self-report scale that measures the severity of fatigue and its effect on a person's activities. The items are scored on a 7-point scale with 1 = strongly disagree and 7= strongly agree, higher scores reflecting more fatigue.
Change in Becks Depression Inventory (BDI) | Assessment at baseline and at week 4, 8, 12, and 16.
  Change in BDI score is studied by comparing baseline value with values at several assessment points throughout the study.
  BDI is a widely used self-report instrument for assessing the degree of depression and changes in depression level. The inventory consists of 21 items about different symptoms and attitudes which are to be valued on a four point scale ranging from 0-3. A total score is calculated by summarizing the scores of the 21 items. Higher total scores indicate more severe depressive symptoms.
Change in SF-36 Health Survey | Assessment at baseline and at week 4, 8, 12, and 16.
  Change in SF-36 score and subscores are studied by comparing baseline values with values at several assessment points throughout the study.
  The SF-36 Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in each section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability, the higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are:
  * vitality
  * physical functioning
  * bodily pain
  * general health perceptions
  * physical role functioning
  * emotional role functioning
  * social role functioning
  * mental health

OTHER OUTCOMES:
Plasma concentrations of OSU6162 | Assessment at week 4 and 16.
  Blood samples are drawn 1-2 h after tablet intake at week 4 and 16, to measure plasma concentrations of OSU6162 after end of study. Plasma concentrations will be analyzed using LC-MS/MS after clinical trial end to ensure blinding. OSU6162 concentrations give an indication of compliance and may be important in studying treatment response.
Adverse Events (AE) or Serious Adverse Events (SAE) - safety assessment | Assessment at baseline and week 2, 4, 6, 8, 10, 12, 14, 16 and 20.
  Patients are asked for the presence of AE/SAE during all visits, both physical visits at the clinic and telephone interviews, throughout the study. Patients are encouraged to make contact with the investigator or study nurse in case of an AE/SAE. AEs are coded using Medical Dictionary for Regulatory Activities (MedDRA) and tabulated by System Organ Class (SOC) and preferred term. All AE/SAE are recorded in the CRF. SAE or SUSAR (suspected unexpected serious adverse event) are immediately reported to the sponsor, CAs, European Medicines Agency and IECs.
Physical and neurological examinations - safety assessment | Assessment at baseline and week 4, 8, 12, 16 and 20.
  Patients undergo standard physical and neurological examinations during all physical visits at the clinic.
Systolic and diastolic blood pressure - safety assessment | Assessment at baseline and week 4, 8, 12, 16 and 20.
  Supine systolic and diastolic blood pressure (mmHg) after lying down for 5 minutes
Heart rate - safety assessment | Assessment at baseline and week 4, 8, 12, 16 and 20.
  Supine heart rate (beats per minute) after lying down for 5 minutes
Electrocardiogram - safety assessment | Assessment at baseline and week 16.
  A standard 12-lead ECG is recorded at baseline and end of treatment (week 16)
Clinical laboratory safety tests | Assessment at baseline and week 4 and 16.
  Blood and urine samples are collected at baseline and week 4 and 16 for analyses of safety blood variables including: clinical chemistry, haematology, urinanalysis, drug screen and pregnancy test.

CONTACTS AND LOCATIONS:
Overall Officials: Carl-Gerhard Gottfries, Prof., Principal Investigator — Gottfries Clinic
Locations (1):
- Gottfries Clinic AB, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EU Clinical Trials Register — http://www.clinicaltrialsregister.eu/ctr-search/trial/2016-003888-19/SE